CLINICAL TRIAL: NCT00674947
Title: A Phase I Study of BIIB015, a Humanized, IgG1, DM4-Conjugated, Anti-Cripto, Monoclonal Antibody, for the Treatment of Subjects With Relapsed or Refractory Solid Tumors
Brief Title: A Phase I Study of BIIB015 in Relapsed/Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Julie Morrissey, Quintiles, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 207ST101
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Solid Tumors
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Recurrence | interventions — huB3F6-SPDB-DM4 immunoconjugate

INTERVENTIONS:
Drug: BIIB015 — IV infusion once every 3 weeks until disease progression or unacceptable toxicity

SUMMARY:
Phase 1, open-labeled, safety and tolerability study for the treatment of subjects with relapsed or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older at the time of informed consent.
* Solid tumors that are relapsed or refractory to at least 1 prior anti-cancer systemic therapy and for which no standard therapy exists.
* ECOG Performance Status </= 2.

Exclusion Criteria

* History of keratoconjunctivitis, open or closed angle glaucoma, or "dry eye" disease.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction within 6 months prior to Day 1.
* Presence of >/= Grade 2 peripheral neuropathy.
* Known presence of central nervous system or brain metastases.
* Prior therapy with a conjugated or unconjugated maytansine derivative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate safety | ongoing
To determine the maximum-tolerated dose (MTD) | ongoing

SECONDARY OUTCOMES:
To evaluate pharmacokinetics (PK) | ongoing
To evaluate clinical activity | ongoing

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Santa Monica, California
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, San Antonio, Texas